CLINICAL TRIAL: NCT00645398
Title: A 13-week, Randomized, Double-Blind, Placebo-Controlled, Monotherapy Trial of Pregabalin (BID) in Patients With Fibromyalgia
Brief Title: A Study of the Efficacy and Safety of Pregabalin for the Treatment of Fibromyalgia
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Pfizer's Upjohn has merged with Mylan to form Viatris Inc. (Industry)
Responsible Party: Sponsor
Organization: Pfizer (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: A0081056
Record Dates: First submitted 2008-03-25; First posted 2008-03-27 (Estimated); Last update posted 2021-01-25 (Actual); Status verified 2008-04

CONDITIONS: Fibromyalgia
MeSH Terms: conditions — Fibromyalgia | interventions — Pregabalin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- A (Experimental)
  Interventions: Drug: Pregabalin
- B (Experimental)
  Interventions: Drug: Pregabalin
- C (Experimental)
  Interventions: Drug: Pregabalin
- D (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Pregabalin — Pregabalin 225 mg BID taken orally, 2 capsules BID for 13 weeks (1 week titration phase + 12 weeks fixed-dose phase).
  Arms: B
Drug: Pregabalin — Pregabalin 150 mg BID taken orally, 2 capsules BID for 13 weeks (1 week titration phase + 12 weeks fixed-dose phase).
  Arms: A
Drug: Pregabalin — Pregabalin 300 mg BID taken orally, 2 capsules BID for 13 weeks (1 week titration phase + 12 weeks fixed-dose phase).
  Arms: C
Drug: Placebo — Matching placebo capsules taken orally, 2 capsules BID for 13 weeks (1 week titration phase + 12 weeks fixed-dose phase).
  Arms: D

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of pregabalin versus placebo for the symptomatic relief of pain associated with fibromyalgia. If this objective is met, then the second objective will be to evaluate the efficacy and safety of pregabalin versus placebo for the management of fibromyalgia (pain, patient global assessment, and functional status). Additionally, the study will evaluate the efficacy of pregabalin versus placebo to improve sleep, fatigue, and mood disturbance associated with fibromyalgia.

ELIGIBILITY:
Inclusion Criteria:

* Patients who met the American College of Rheumatology (ACR) criteria for fibromyalgia (ie, widespread pain present for at least 3 months, and pain in at least 11 of 18 specific tender point sites)
* Patients who completed at least 4 pain diaries within the last 7 days and the average pain score must have been ≥4, and had a score of ≥40 mm on the Visual Analogue Scale (VAS) of the SF-MPQ at screening (Visit 1) and randomization (Visit 2)

Exclusion Criteria:

* Patients with other severe pain that may confound assessment or self-evaluation of the pain associated with fibromyalgia
* Patients with any inflammatory muscle or rheumatologic disease other than fibromyalgia, active infections, or untreated endocrine disorders
* Patients with severe depression

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 751 (Actual)
Dates: Start 2004-09; Study Completion 2005-06 (Actual)

PRIMARY OUTCOMES:
Endpoint mean pain score derived from the subject's daily pain diary | Endpoint
Patient Global Assessment (Patient Global Impression of Change) at Termination Visit | Weeks 5 and 13
Change from baseline in functioning (score created from the Short Form-36 [SF-36] Social and Physical Functioning, Fibromyalgia Impact Questionnaire [FIQ]-Total Score, and Sheehan Disability Scale [SDS] Total Score) at Termination Visit | Baseline and Weeks 5, 9, and 13

SECONDARY OUTCOMES:
Change from baseline in FIQ scores at Weeks 5, 9, and 13 | Baseline and Weeks 5, 9, and 13
Change from baseline in SDS scores at Weeks 5, 9, and 13 | Baseline and Weeks 5, 9, and 13
Change from baseline in Medical Outcomes Study (MOS)-Sleep Scale scores at Weeks 5, 9, and 13 | Baseline and Weeks 5, 9, and 13
Quality of Sleep Score from the Daily Sleep Diary | Daily
Change from baseline in Multidimensional Assessment of Fatigue (MAF) scores at Weeks 5, 9, and 13 | Baseline and Weeks 5, 9, and 13
Change from baseline in Hospital Anxiety and Depression Scale (HADS) scores at Week 13 | Baseline and Week 13
Change from baseline in Short Form McGill Pain Questionnaire (SF-MPQ) scores at Weeks 5, 9, and 13 | Screening, baseline, and Weeks 5, 9, and 13
Change from baseline in Fibromyalgia Health Assessment Questionnaire (F-HAQ) scores at Weeks 9 and 13 | Baseline and Weeks 9 and 13
Adverse events | Weeks 1, 2, 5, 9, 13, and at follow-up
Physical examination, including vital signs and weight | Baseline and Week 5 (vital signs only) and 13
Neurological examination | Screening and Week 13
Electrocardiogram | Screening and Week 13
Laboratory tests, including chemistry and hematology | Baseline and Weeks 5, 13, and at follow-up
Urinalysis | Baseline and Weeks 13 and at follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (84):
- United States (84):
  - Pfizer Investigational Site, Birmingham, Alabama
  - Pfizer Investigational Site, Huntsville, Alabama
  - Pfizer Investigational Site, Paradise Valley, Arizona
  - Pfizer Investigational Site, Phoenix, Arizona
  - Pfizer Investigational Site, Scottsdale, Arizona
  - Pfizer Investigational Site, Hot Springs, Arkansas
  - Pfizer Investigational Site, Little Rock, Arkansas
  - Pfizer Investigational Site, Beverly Hills, California
  - Pfizer Investigational Site, Long Beach, California
  - Pfizer Investigational Site, Los Alamitos, California
  - Pfizer Investigational Site, Newport Beach, California
  - Pfizer Investigational Site, Northridge, California
  - Pfizer Investigational Site, Pismo Beach, California
  - Pfizer Investigational Site, Redondo Beach, California
  - Pfizer Investigational Site, Riverside, California
  - Pfizer Investigational Site, Walnut Creek, California
  - Pfizer Investigational Site, Whittier, California
  - Pfizer Investigational Site, Danbury, Connecticut
  - Pfizer Investigational Site, New Milford, Connecticut
  - Pfizer Investigational Site, Stratford, Connecticut
  - Pfizer Investigational Site, Clearwater, Florida
  - Pfizer Investigational Site, Miami, Florida
  - Pfizer Investigational Site, Ocala, Florida
  - Pfizer Investigational Site, Palm Beach Gardens, Florida
  - Pfizer Investigational Site, Plantation, Florida
  - Pfizer Investigational Site, St. Petersburg, Florida
  - Pfizer Investigational Site, Sunrise, Florida
  - Pfizer Investigational Site, West Palm Beach, Florida
  - Pfizer Investigational Site, Atlanta, Georgia
  - Pfizer Investigational Site, Decatur, Georgia
  - Pfizer Investigational Site, Boise, Idaho
  - Pfizer Investigational Site, Chicago, Illinois
  - Pfizer Investigational Site, Maywood, Illinois
  - Pfizer Investigational Site, Oak Brook, Illinois
  - Pfizer Investigational Site, Peoria, Illinois
  - Pfizer Investigational Site, Kansas City, Kansas
  - Pfizer Investigational Site, Overland Park, Kansas
  - Pfizer Investigational Site, Madisonville, Kentucky
  - Pfizer Investigational Site, New Orleans, Louisiana
  - Pfizer Investigational Site, Newton, Massachusetts
  - Pfizer Investigational Site, East Lansing, Michigan
  - Pfizer Investigational Site, Kalamazoo, Michigan
  - Pfizer Investigational Site, Lansing, Michigan
  - Pfizer Investigational Site, Kansas City, Missouri
  - Pfizer Investigational Site, Lebanon, New Hampshire
  - Pfizer Investigational Site, Princeton, New Jersey
  - Pfizer Investigational Site, Albany, New York
  - Pfizer Investigational Site, New York, New York
  - Pfizer Investigational Site, Rochester, New York
  - Pfizer Investigational Site, Charlotte, North Carolina
  - Pfizer Investigational Site, Wilmington, North Carolina
  - Pfizer Investigational Site, Winston-Salem, North Carolina
  - Pfizer Investigational Site, Cincinnati, Ohio
  - Pfizer Investigational Site, Columbus, Ohio
  - Pfizer Investigational Site, Mogadore, Ohio
  - Pfizer Investigational Site, Toledo, Ohio
  - Pfizer Investigational Site, Oklahoma City, Oklahoma
  - Pfizer Investigational Site, Eugene, Oregon
  - Pfizer Investigational Site, Medford, Oregon
  - Pfizer Investigational Site, Portland, Oregon
  - Pfizer Investigational Site, Altoona, Pennsylvania
  - Pfizer Investigational Site, Duncansville, Pennsylvania
  - Pfizer Investigational Site, Johnstown, Pennsylvania
  - Pfizer Investigational Site, Mechanicsburg, Pennsylvania
  - Pfizer Investigational Site, Philadelphia, Pennsylvania
  - Pfizer Investigational Site, Pittsburgh, Pennsylvania
  - Pfizer Investigational Site, Pottstown, Pennsylvania
  - Pfizer Investigational Site, West Reading, Pennsylvania
  - Pfizer Investigational Site, Wyomissing, Pennsylvania
  - Pfizer Investigational Site, Anderson, South Carolina
  - Pfizer Investigational Site, Charleston, South Carolina
  - Pfizer Investigational Site, Greer, South Carolina
  - Pfizer Investigational Site, Memphis, Tennessee
  - Pfizer Investigational Site, Nashville, Tennessee
  - Pfizer Investigational Site, Austin, Texas
  - Pfizer Investigational Site, Dallas, Texas
  - Pfizer Investigational Site, Lubbock, Texas
  - Pfizer Investigational Site, Richardson, Texas
  - Pfizer Investigational Site, San Antonio, Texas
  - Pfizer Investigational Site, Salt Lake City, Utah
  - Pfizer Investigational Site, Woodstock, Vermont
  - Pfizer Investigational Site, Virginia Beach, Virginia
  - Pfizer Investigational Site, Seattle, Washington
  - Pfizer Investigational Site, Yakima, Washington

REFERENCES:
- [Derived] Clair A, Emir B. The safety and efficacy of pregabalin for treating subjects with fibromyalgia and moderate or severe baseline widespread pain. Curr Med Res Opin. 2016;32(3):601-9. doi: 10.1185/03007995.2015.1134463. Epub 2016 Jan 27. PMID 26694975
- [Derived] Straube S, Moore RA, Paine J, Derry S, Phillips CJ, Hallier E, McQuay HJ. Interference with work in fibromyalgia: effect of treatment with pregabalin and relation to pain response. BMC Musculoskelet Disord. 2011 Jun 3;12:125. doi: 10.1186/1471-2474-12-125. PMID 21639874
- [Derived] Bhadra P, Petersel D. Medical conditions in fibromyalgia patients and their relationship to pregabalin efficacy: pooled analysis of Phase III clinical trials. Expert Opin Pharmacother. 2010 Dec;11(17):2805-12. doi: 10.1517/14656566.2010.525217. Epub 2010 Nov 2. PMID 21039311
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A0081056&StudyName=A%20Study%20of%20the%20Efficacy%20and%20Safety%20of%20Pregabalin%20for%20the%20Treatment%20of%20Fibromyalgia